CLINICAL TRIAL: NCT07151066
Title: Examination of the Relationship Between the Anthropometric Parameters of the Foot and Plantar Fasciitis
Brief Title: Anthropometric Parameters of the Foot and Plantar Fasciitis
Acronym: PF
Status: Enrolling by invitation | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Hande YAZICI, Lecturer, Medipol University
Other Study IDs: E-10840098-202.3.02-5582
Record Dates: First submitted 2025-08-27; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Plantar Fasciitis
Keywords: Foot anthropometric measurements; Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PF Group: individuals with plantar fasciitis

SUMMARY:
The aim of this study is to systematically evaluate anthropometric and lifestyle parameters in individuals diagnosed with PF and compare them with healthy individuals. This will reveal the structural and behavioural risk factors involved in the development of PF, providing a scientific basis for preventive measures and orthotic approaches.

Assessment Parameters:

Medical History Form

1. Demographic data: Age, height, weight, BMI
2. Foot anthropometric measurements
3. Footwear preference: Footwear Assessment Score ( Footwear Assessment Score )
4. Lower extremity joint health: History of pain, injury, or limitation in the knee and hip joints
5. Daily step count: Measurement using the Step Counter mobile application
6. Physical activity level: IPAQ-SF (International Physical Activity Questionnaire - Short Form) questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 65 years of age,
* Having been diagnosed with plantar fasciitis,
* Having heel pain complaints originating from the plantar medial calcaneal tubercle,
* Pain complaints being most pronounced in the first steps taken in the morning or after rest,

Exclusion Criteria:

* Any cardiopulmonary, dermatological, neurological or orthopaedic problems,
* History of lower limb surgery,
* Use of assistive devices (walker, crutches, etc.)
* Cognitive, mental and/or psychological problems
* Pregnancy
* Lower limb amputation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with plantar fasciitis by the Orthopaedics and Traumatology Department at Medipol Hospital
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Anthropometric measurements of the foot | baseline
  * Foot length
  * Metatarsal width
  * Medial arch height

CONTACTS AND LOCATIONS:
Overall Officials: Naile Hande İŞÇİ, PhD (c), Study Chair — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No